CLINICAL TRIAL: NCT04803370
Title: Study of the Efficacy of Reinforcing of the Standard Therapy in COVID-19 Patients With Repeated Transfusion of Immune Plasma From COVID-19 Convalescents vs Exclusive Standard Therapy in Hospitalized COVID-19 Patients
Brief Title: Efficacy of Reinforcing Standard Therapy in COVID-19 Patients With Repeated Transfusion of Convalescent Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Son Llatzer (Other)
Collaborators: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Principal Investigator, Maria Arrizabalaga Asenjo, Principal Investigator, Hospital Son Llatzer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-PLASMA-2020
Record Dates: First submitted 2021-03-09; First posted 2021-03-17 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Covid19
Keywords: COVID19, Immune Plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Other): Standard treatment for COVID-19 (according to clinical guidelines for COVID-19).
  Interventions: Other: Standard treatment for COVID-19
- Intervention group (Experimental): Convalescent patient plasma 300 ml given in 2 consecutive days, plus standard treatment for COVID-19 (according to clinical guidelines).
  Interventions: Other: Convalescent Plasma with antibody against SARS-CoV-2.

INTERVENTIONS:
Other: Convalescent Plasma with antibody against SARS-CoV-2. — Convalescent plasma plus standard treatment for COVID-19. The convalescent plasma is from patients recovered from COVID-19 and negative viremia in the test detection COVID-19.
  The infusions will be given on days 1 and 2, of the study, after the positive result for COVID-19 of the recipient patient.
  Arms: Intervention group
Other: Standard treatment for COVID-19 — The patients will receive the standard treatment for COVID-19, according to guidelines for COVID-19 (retrovirals drugs, interferon-α / β, anti-Interleukin-6 monoclonal antibody, oxygen therapy, etc..)
  Arms: Control group

SUMMARY:
The coronavirus disease 2019 (COVID-19) was classified as a pandemic by the World Health Organization (WHO) in March 2020. The SARS-COV-2 virus is easily transmissible and there is currently no approved treatment with effective results. Although the main epidemiological parameters are currently being studied, apparently the speed of contagion, the incidence and the mortality rate in severe cases appear to be high. Therefore, there is an urgent need to find a viable therapeutic option. The present trial is a pilot study with an objective to determine the efficacy of standard treatment reinforced with two repeated doses in two consecutive days of plasma from former convalescent people of the COVID-19 disease already discharged and / or with results in negative COVID-19 screenings, transfused to hospitalized COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the HIP and sign the study IC
* male or female =/> 18 years
* Patient hospitalized with a COVID-19 diagnosis by PCR on nasopharyngeal swabs or any other biological sample.
* Presence of respiratory symptoms and / or fever associated with COVID-19, with clinical evolution time for COVID-19 equal to or less than 7 days.
* Presence of pneumonia on chest X-ray and / or SatO2 <94% aa.
* Sequential Organ Failure Assessment (SOFA) score ≤ 6.
* Accept the condition of complying with the procedures established in the protocol.

Exclusion Criteria:

* Patients with a previous history of allergic transfusion reaction.
* Lactating or pregnant women and a positive pregnancy test.
* Patients who have been treated with plasma in the 21 days prior to the screening / baseline visit.
* Patients who are at the time of study, participating in another clinical trial.
* Patients who haven't completed all study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Son Llatzer, Palma de Mallorca, Islas de Balears, Spain

REFERENCES:
- [Result] Bargay-Lleonart J, Sarubbo F, Arrizabalaga M, Guerra JM, Borras J, El Haji K, Flexas M, Perales J, Fernandez-Baca V, Gallegos C, Cruz MR, Velasco S, Lopez V, Cruz A, Bautista-Gili A, Jimenez-Marco T, Girona-Llobera E, Vilaplana L, Calonge L, Tena J, Galan MP, Payeras A. Reinforcement of the Standard Therapy with Two Infusions of Convalescent Plasma for Patients with COVID-19: A Randomized Clinical Trial. J Clin Med. 2022 May 27;11(11):3039. doi: 10.3390/jcm11113039. PMID 35683427

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Standard treatment for COVID-19 (according to clinical guidelines for COVID-19).
  Standard treatment for COVID-19: The patients will receive the standard treatment for COVID-19, according to guidelines for COVID-19 (retrovirals drugs, interferon-α / β, anti-IL-6 monoclonal antibody, oxygen therapy, etc..)
- Intervention Group: Convalescent patient plasma 300 ml given in 2 consecutive days, plus standard treatment for COVID-19 (according to clinical guidelines).
  Convalescent Plasma with antibody against SARS-CoV-2.: Convalescent plasma plus standard treatment for COVID-19. The convalescent plasma is from patients recovered from COVID-19 and negative viremia in the test detection COVID-19.
  The infusions will be given on days 1 and 2, of the study, after the positive result for COVID-19 of the recipient patient.
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 17 | 38
Completed | 17 | 37
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 17 | 37 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (3) | 58 (2) | 58 (1.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 21
  Male | 10 | 23 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.34 (1.99) | 30.72 (1.24) | 30.62 (1.05)
Concomitant illnesses [Count of Participants; unit: Participants] — Type of concomitant illnesses are cardiac diseases, respiratory diseases, digestive diseases, neurological diseases, psychiatric diseases, nephrological diseases, ophthalmological diseases, dermatological diseases, endocrinological diseases, rheumatic/osteoarticular diseases and immunity diseases
  Participants
    Yes | 14 | 27 | 41
    No | 3 | 10 | 13
Concomitant medication [Count of Participants; unit: Participants]
  Yes | 7 | 17 | 24
  No | 10 | 20 | 30
Smoke [Count of Participants; unit: Participants]
  Yes | 1 | 2 | 3
  No | 16 | 35 | 51
Drug abuse habits [Count of Participants; unit: Participants] — Addictive use of psychoactive substances such as amphetamines, cocaine, marijuana, ecstasy, etc...
  Participants
    Yes | 1 | 2 | 3
    No | 16 | 35 | 51
Standard treatment [Number; unit: participants]
  Antiinflammatory | 11 | 29 | 40
  Antiviral | 5 | 14 | 19
  Antibiotic | 3 | 10 | 13
  Anticoagulant | 5 | 13 | 18
  Oxygen therapy | 10 | 19 | 29

OUTCOME MEASURES:

1. Primary Outcome: Adaptive COVID-19 Treatment Trial Scale (ACTT) Version II
Description: The scale provides a measure of COVID-19 severity based on the patient's physical situation, whose design was based on a blueprint of the WHO in treating COVID-19.
  * 1= Death
  * 2= Hospitalized. on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  * 3= Hospitalized. on non-invasive ventilation or high flow oxygen devices
  * 4= Hospitalized. requiring supplemental oxygen
  * 5= Hospitalized. not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  * 6= Hospitalized. not requiring supplemental oxygen - no longer requiring ongoing medical care.
  * 7= Not hospitalized. limitation on activities and/or requiring home oxygen
  * 8= Not hospitalized. no limitations on activities.
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
Participants
  Grade 1 | 0 | 0
  Grade 2 | 0 | 0
  Grade 3 | 2 | 3
  Grade 4 | 5 | 6
  Grade 5 | 4 | 10
  Grade 6 | 2 | 3
  Grade 7 | 1 | 3
  Grade 8 | 3 | 12

2. Primary Outcome: Adaptive COVID-19 Treatment Trial Scale (ACTT) Version II
Description: as for outcome 1
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
Participants
  Grade 1 | 0 | 0
  Grade 2 | 1 | 0
  Grade 3 | 0 | 2
  Grade 4 | 1 | 2
  Grade 5 | 1 | 3
  Grade 6 | 3 | 3
  Grade 7 | 5 | 9
  Grade 8 | 6 | 18

3. Secondary Outcome: Anti-SARS-CoV-2 S IgG Serum Titer
Description: The levels of Anti-SARS-CoV-2 S IgG serum
Time Frame: At inclusion, Day 21
Measure: Mean (Standard Error); unit: AU/ ml
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
AU/ ml
  At inclusion | 90.28 (53.51) | 98.16 (39.89)
  Day 21 | 773.84 (327.53) | 1102.81 (194.51)

4. Secondary Outcome: Time of Hospitalization
Description: time that the patients have passed in the hospital.
Time Frame: Day 21
Measure: Mean (Standard Error); unit: days
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
days | 10.5 (1.8) | 8.9 (0.9)

5. Secondary Outcome: Time to Negativization of RT-PCR
Description: total time elapsed until negative RT-PCR test
Time Frame: Day 21
Measure: Mean (Standard Error); unit: days
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
days | 14.6 (2.1) | 12.4 (1.4)

6. Secondary Outcome: Diastolic Blood Pressure
Description: the pressure of blood in the artery when the heart relaxes between beats.
Time Frame: At inclusion, Day 1, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
mmHg
  At inclusion | 79.62 (3.17) | 75.21 (2.12)
  Day 1 | 77.18 (5.01) | 74.83 (1.72)
  Day 3 | 75.25 (2.84) | 74.33 (2.08)
  Day 7 | 81.07 (3.53) | 72.48 (1.38)
  Day 14 | 80.72 (5.06) | 78.96 (1.71)
  Day 21 | 83.83 (3.91) | 81.85 (1.82)

7. Secondary Outcome: Systolic Blood Pressure
Description: The pressure of blood in the artery when the heart contracts. It is the high number in a blood pressure measurement.
Time Frame: At inclusion, Day 1, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
mmHg
  At inclusion | 130.62 (5.84) | 121.11 (3.25)
  Day 1 | 135 (7.53) | 123.87 (3.25)
  Day 3 | 134.2 (3.34) | 121.94 (2.15)
  Day 7 | 141.53 (6.85) | 119.48 (2.82)
  Day 14 | 145.8 (6.57) | 125.77 (2.56)
  Day 21 | 145.81 (6.01) | 128.39 (2.84)

8. Secondary Outcome: Temperature
Time Frame: At inclusion, Day 1, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: degrees Celsius
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
degrees Celsius
  At inclusion | 36.79 (0.26) | 36.43 (0.14)
  Day 1 | 36.59 (0.14) | 36.48 (0.09)
  Day 3 | 36.61 (0.19) | 36.50 (0.11)
  Day 7 | 36.24 (0.17) | 36.17 (0.09)
  Day 14 | 36.58 (0.18) | 36.46 (0.10)
  Day 21 | 36.26 (0.10) | 36.38 (0.10)

9. Secondary Outcome: Cardiac Frequency
Description: The number of heart contractions or beats per unit of time. The normal values in adults at rest range between 60 and 100 beats per minit.
Time Frame: At inclusion, Day 1, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: beats/minit
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
beats/minit
  At inclusion | 83.37 (4.05) | 79.82 (2.25)
  Day 1 | 75.54 (4.08) | 79.57 (2.34)
  Day 3 | 77.31 (3.16) | 73.73 (2.10)
  Day 7 | 79.77 (4.28) | 68.35 (2.24)
  Day 14 | 86.27 (5.71) | 85.38 (2.66)
  Day 21 | 84.90 (5.31) | 86.72 (3.01)

10. Secondary Outcome: Respiratory Frequency
Description: Number of breaths the patient takes per minute.
Time Frame: At inclusion, Day 1, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: breath/minut
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
breath/minut
  At inclusion | 20.06 (1.27) | 22.42 (1.25)
  Day 1 | 22.36 (1.20) | 23.61 (1.13)
  Day 3 | 20.23 (0.92) | 22.65 (0.98)
  Day 7 | 21.12 (1.29) | 19.95 (1.05)
  Day 14 | 18.16 (1.27) | 18.42 (0.66)
  Day 21 | 16.43 (0.61) | 19.38 (1.11)

11. Secondary Outcome: Oxygen Saturation
Description: blood oxygen percentage. A healthy percentage of oxygen in the blood is between 95% and 100%.
Time Frame: At inclusion, Day 1, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: percentage of blood oxygen
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
percentage of blood oxygen
  At inclusion | 95.31 (0.73) | 95.4 (0.42)
  Day 1 | 95.63 (0.67) | 95.21 (0.94)
  Day 3 | 95.18 (0.51) | 95.78 (0.38)
  Day 7 | 94.69 (0.82) | 95.82 (0.42)
  Day 14 | 95.1 (0.54) | 95.73 (0.43)
  Day 21 | 96 (0.52) | 96.15 (0.37)

12. Secondary Outcome: Hemoglobin
Description: hemoglobin levels in the blood
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
g/dL
  At inclusion | 13.38 (0.31) | 13.45 (0.29)
  Day 3 | 13.05 (0.34) | 12.83 (0.31)
  Day 7 | 12.98 (0.37) | 13.21 (0.35)
  Day 14 | 12.94 (0.31) | 13.37 (0.28)
  Day 21 | 12.51 (0.4) | 13.04 (0.37)

13. Secondary Outcome: Leucocytes
Description: Leucocyte count a patient's blood.
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: cells x10^9/L
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
cells x10^9/L
  At inclusion | 7.81 (0.87) | 7.40 (0.46)
  Day 3 | 8.31 (0.90) | 8.67 (0.65)
  Day 7 | 10.43 (0.87) | 9.97 (0.66)
  Day 14 | 9.32 (1.08) | 9.40 (0.82)
  Day 21 | 6.47 (0.61) | 6.20 (0.45)

14. Secondary Outcome: Neutrophils
Description: Neutrophils count a patient's blood.
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: cells x10^9/L
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
cells x10^9/L
  At inclusion | 6.11 (0.86) | 5.50 (0.48)
  Day 3 | 6.27 (0.85) | 6.37 (0.61)
  Day 7 | 7.60 (0.78) | 6.75 (0.68)
  Day 14 | 6.53 (1.16) | 6.58 (0.83)
  Day 21 | 4.17 (0.59) | 3.74 (0.40)

15. Secondary Outcome: Absolute Lymphocytes
Description: lymphocyte count a patient's blood.
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: cells x10^9/L
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
cells x10^9/L
  At inclusion | 1.165 (0.11) | 1.44 (0.15)
  Day 3 | 1.32 (0.17) | 1.36 (0.10)
  Day 7 | 1.94 (0.26) | 2.07 (0.16)
  Day 14 | 2.02 (0.21) | 2.14 (0.15)
  Day 21 | 1.63 (0.18) | 1.88 (0.12)

16. Secondary Outcome: Activated Partial Thromboplastin Time
Description: measurement of the number of seconds it takes for a clot to form in a patient's blood.
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
seconds
  At inclusion | 29.62 (1.43) | 30.62 (0.70)
  Day 3 | 27.96 (0.64) | 29.62 (0.76)
  Day 7 | 27.49 (0.62) | 28.72 (0.73)
  Day 14 | 28.29 (0.88) | 29.37 (0.67)
  Day 21 | 31.39 (2.03) | 31.12 (0.73)

17. Secondary Outcome: Fibrinogen Level
Description: measurement of the level of fibrinogen in the blood (mg / dl), as a measure of assessing the severity of the disease.
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
mg/dL
  At inclusion | 713.13 (44.64) | 732.36 (32.57)
  Day 3 | 671.94 (42.38) | 683.43 (33.11)
  Day 7 | 591.44 (36.40) | 559.77 (32.01)
  Day 14 | 562.67 (38.92) | 531.46 (35.71)
  Day 21 | 527.23 (39.46) | 511.96 (33.35)

18. Secondary Outcome: Fragment D-dimer Assessment
Description: Determination of the existence of the D-dimer fragment in blood as a measure of assessing the severity of the disease.
Time Frame: At inclusion, Day 3, Day 7, Day 14
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
ng/mL
  At inclusion | 350.26 (62.80) | 294.11 (36.63)
  Day 3 | 443.2 (77.12) | 377.52 (117.12)
  Day 7 | 321.63 (61.81) | 377.03 (91.58)
  Day 14 | 300.69 (51.74) | 222.8 (24.66)

19. Secondary Outcome: Glomerular Filtration Rate Assessment
Description: estimation of how much blood passes per minute through the glomerular filters of the kidneys (ml/min).
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: ml/min
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
ml/min
  At inclusion | 80.44 (5.41) | 93.65 (3.31)
  Day 3 | 86.15 (4.07) | 96.68 (3.35)
  Day 7 | 87.04 (4.60) | 96.81 (3.55)
  Day 14 | 80.17 (5.29) | 92.24 (3.35)
  Day 21 | 83.98 (4.59) | 92.53 (3.71)

20. Secondary Outcome: Troponin I Assessment
Description: measurement of the levels of troponin I proteins in the blood (ng/mL), as a measure of assessing the severity of the disease.
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
ng/mL
  At inclusion | 6.55 (1.59) | 5.45 (0.65)
  Day 3 | 5.86 (1.57) | 6.41 (0.78)
  Day 7 | 5.50 (1.56) | 6.14 (1.10)
  Day 14 | 5.24 (1.80) | 4.32 (0.57)
  Day 21 | 5.44 (1.27) | 4.24 (0.56)

21. Secondary Outcome: Procalcitonin Assessment
Description: measurement of the levels of procalcitonin in the blood (ng/L), as a measure of assessing the severity of the disease.
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: ng/L
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
ng/L
  At inclusion | 0.86 (0.73) | 0.11 (0.02)
  Day 3 | 0.78 (0.70) | 0.09 (0.02)
  Day 7 | 0.44 (0.39) | 0.05 (0.01)
  Day 14 | 0.04 (0.005) | 0.04 (0.004)
  Day 21 | 0.05 (0.01) | 0.04 (0.01)

22. Secondary Outcome: C-reactive Protein Assessment
Description: measurement of the level of c-reactive protein in the blood (mg/dl), as a measure of a change in inflammation
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
mg/dL
  At inclusion | 64.19 (15.81) | 55.39 (9.20)
  Day 3 | 52.25 (12.77) | 43.51 (8.67)
  Day 7 | 33.83 (11.42) | 16.60 (3.55)
  Day 14 | 18.49 (4.85) | 9.18 (1.97)
  Day 21 | 17.46 (5.35) | 8.72 (1.72)

23. Secondary Outcome: Lactate Dehydrogenase (LDH) Assessment
Description: measurement of the level of lactate dehydrogenase in the blood (U/L), as a measure of assessing the severity of the disease.
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: Unit/L
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
Unit/L
  At inclusion | 283.56 (12.78) | 306.31 (21.80)
  Day 3 | 286.47 (15.27) | 317.18 (25.14)
  Day 7 | 276.67 (17.50) | 267.6 (16.95)
  Day 14 | 277 (27.41) | 232.25 (9.21)
  Day 21 | 246.38 (21.33) | 215.04 (8.10)

24. Secondary Outcome: Interleukin-6 Assessment
Description: measurement of serum levels Interleukin-6 in pg/mL, as a measure of assessing the severity of the disease.
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
pg/mL
  At inclusion | 29.48 (6.01) | 32.60 (5.21)
  Day 3 | 28.18 (4.10) | 25.37 (5.83)
  Day 7 | 17.33 (3.54) | 12.24 (3.12)
  Day 14 | 11.31 (3.45) | 12.02 (2.53)
  Day 21 | 10.76 (2.68) | 11.80 (3.31)

25. Secondary Outcome: Ferritin Blood Assessment
Description: measurement of the amount of ferritin (blood protein) in ng/ml in the blood, as a measure of assessing the severity of the disease.
Time Frame: At inclusion, Day 3, Day 7, Day 14, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
ng/mL
  At inclusion | 566.48 (158.23) | 745.60 (129.99)
  Day 3 | 626.24 (136.86) | 736.80 (119.52)
  Day 7 | 624.35 (124.99) | 670.25 (92.21)
  Day 14 | 412.88 (78.48) | 450.42 (60.09)
  Day 21 | 392.57 (123.70) | 272.27 (48.16)

26. Secondary Outcome: Percentage of Patients Requiring Admission to Intensive Care Units.
Description: Percentage of patients requiring admission to intensive care units.
Time Frame: Day 21
Measure: Number; unit: percentage of participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
percentage of participants
  yes | 16 | 17
  No | 84 | 83

27. Secondary Outcome: Mortality Rate at 15 Days
Description: number of dead participants through day 15
Time Frame: Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
Participants | 0 | 0

28. Secondary Outcome: Mortality Rate at 30 Days
Description: number of dead participants through day 30
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 37
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 days
Description: [Not Specified]
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/37
Other Adverse Events (participants affected / at risk) | 0/17 | 4/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=17) | Intervention Group (N=37)
Skin rash (Grade 1) (Skin and subcutaneous tissue disorders) | 0 | 1
Left ear hearing los (Ear and labyrinth disorders) | 0 | 1
Mild dizziness (Nervous system disorders) | 0 | 1
Left hypochondrium pain (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT04803370/Prot_SAP_ICF_000.pdf